CLINICAL TRIAL: NCT02543385
Title: The Use of S Ketamine Versus Placebo During Target Controlled Intravenous Anaesthesia to Reduce Morphine Consumption and Side-Effects After Abdominal Hysterectomy: A Randomized Control Trial
Brief Title: S Ketamine Use in Total Abdominal Hysterectomy
Acronym: SKET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of protocol title
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008/905/D
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Total Abdominal Hysterectomy
Keywords: S Ketamine; Morphine; Consumption
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKET (Active Comparator): Intravenous S+ketamine 0.25 mg/kg (i.v. bolus) at the beginning and 0.25 mg/kg (i.v. bolus) 20 minutes before extubation along with remifentanil according to Minto model and propofol infusion according to Schnider model through target control infusion pump.
  Interventions: Drug: S Ketamine
- PLACEBO (Placebo Comparator): Intravenous normal saline (as placebo, with similar volume) at the beginning and 20 minutes before extubation along with remifentanil according to Minto model and propofol according to Schnider model through target control infusion pump.
  Interventions: Drug: S Ketamine

INTERVENTIONS:
Drug: S Ketamine — S+ketamine will be given in group I only in the doses of 0.25mg/kg (iv bolus) before induction along with midazolam and 0. 25 mg/kg (iv bolus) 20 minutes prior to extubation

SUMMARY:
This study investigates the effect of low dose S+ketamine compared to placebo on cumulative morphine consumption at 24 hours in women undergoing open abdominal hysterectomy with remifentanil-propofol target controlled infusion. It compares the adverse effect profile in patients receiving S+ketamine as compared to those who did not. Participants are randomly distributed in two groups of 45 patient's each.

DETAILED DESCRIPTION:
In recent times it has been suggested that NMDA receptor antagonist like ketamine when used in small doses helps reducing postoperative pain and opioid consumption without compromising wakefulness and or causing its psycho mimetic adverse effect .

The clinical utility of S+ ketamine as an adjuvant intra-operatively remains controversial. The NMDA receptor activation and subsequent biochemical process has been proven to play an important role in both hyperalgesia after tissue injury and the development of opioid tolerance. Various studies have reported the advantage of S+ ketamine over traditional balanced anaesthesia, but may lead to secondary hyperalgesia and increased opioid requirement in post operative period in both animals and healthy human volunteers. Other studies showed that 48 hours continuous administration of small-dose ketamine, together with patient-controlled analgesia (PCA) with morphine, or systemic, epidural co-administration of ketamine and opiates markedly reduced cumulative morphine. However, the dosage, route and timing of administration of S+-ketamine varied in different setting.

ELIGIBILITY:
Inclusion Criteria:

* Females above the age of 21 years old scheduled undergoing open abdominal hysterectomy with remifentanil-propofol TCI in KKH for benign condition (fibroids, adenomyosis),
* Be willing and able to give written informed consent for participation in this study
* ASA I/II patient's.

Exclusion Criteria:

* Patient with contraindications to the use of S+ketamine, as listed in the product label e.g. untreated or insufficiently treated thyroid hyperfunction, unstable angina pectoris or myocardial infarction within the last 6 months, diseases of the CNS, increased intraocular pressure and perforating ocular injuries, surgical procedures in the upper respiratory tract, etc
* Patients with a h/o drug or alcohol abuse
* Regular use of analgesics, or use of opioids within 12 hours of surgery
* Patient on chronic use of benzodiazepine or neurololeptics
* Patient on thyroid replacement hormone
* H/o IHD,HTN,Thyroid disorder.
* BMI> 30kg/m2.
* H/o Psychiatric disorder.
* Laproscopic surgery converted to open surgery.
* Pregnant or breast feeding female's.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
S ketamine used in TAH | 1 YEAR